CLINICAL TRIAL: NCT06680362
Title: Anatomical Characteristics of the Splenic Artery in Northwest China and Its Impact on Laparoscopic Radical Total Gastrectomy
Brief Title: The Influence of Splenic Artery Characteristics in Gastric Cancer Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: xiaohua li (Other)
Responsible Party: Sponsor-Investigator, xiaohua li, professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Other Study IDs: KY20242177-C-1
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Gastrectomy; Gastric Carcinoma
Keywords: Gastric carcinoma; Hilus lienis; Vascular anatomy; Ethnicity
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — As the study is observational, no specific samples should be collected. It is only necessary to collect the anatomic characteristics and perioperative data of the splenic artery in the included population
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concentrated group: If the distance between the bifurcation of the splenic artery and the splenic hilum was less than 2 cm, the patient was assigned to the concentrated group
- distributed group: If the distance between the splenic artery bifurcation and the splenic portal is greater than or equal to 2cm, it is classified as distributed group

SUMMARY:
The northwest Chinese population has unique anatomical characteristics of splenic artery due to ethnic differences, which has an important impact on the development and prognosis of laparoscopic radical total gastrectomy.

DETAILED DESCRIPTION:
Gastric carcinoma (GC) is the fifth most common malignancy and the fourth most common cause of cancer death worldwide, which has severely affected human health. Although a variety of combined treatment methods, such as chemotherapy and immunotherapy, have improved the treatment effect in recent years, surgery is still the only curative option. The latest CSCO guidelines recommend that splenic hilar lymph nodes must be dissected during total gastrectomy combined with D2 lymph node dissection for advanced gastric cancer. However, as a result of the deep position of the splenic hilum, complicated and variant vessels and covered with fascial tissue, it is difficult to dissect the lymph nodes in the upper pancreatic and splenic hilum regions, which increases the risk of surgery and the difficulty of prognosis recovery. Therefore, a more complete classification and summary of the characteristics of splenic artery will assure the evaluation and implementation of radical gastrectomy.

Currently, a wide variety of classification criteria apply to splenic arteries. One study reported that the splenic artery can be divided into superficial, middle and concealed, based on its location relative to the pancreas. Splenic artery trajectories can also be classified as straight, sinusoidal, serpentine, or alternating. Particularly, it is widely accepted that Zheng et al.'s anatomical classification and clinical implications of the splenic artery are more in-depth and comprehensive. The splenic artery was classified according to the number of branches of its secondary vessels, its position relative to the pancreas, and the distance of the terminal end of the main trunk from the splenic hilum. The results of this study, which focused mainly on the southeastern population, revealed differences in the impact of splenic artery classification on surgery. However, due to different races and the anatomical structure, the classification of the splenic artery differed, which in turn affects the operation and prognosis. In contrast to the study of Zheng et al., which focused primarily on a population in Southeast China, the differences in the anatomical characteristics of the splenic artery in the population in Northwest China may have different effects on the development and prognosis of laparoscopic radical total gastrectomy.

Therefore, we conducted this study to analyze and summarize the characteristics of splenic artery classification and its impact on laparoscopic radical total gastrectomy in the northwest Chinese population.

Inpatients who underwent laparoscopic radical total gastrectomy at the Department of Gastrointestinal Surgery of the First Affiliated Hospital of Air Force Medical University were enrolled. All patients were recruited from five provinces in Northwest China, including Shaanxi Province, Gansu Province, Qinghai Province, the Ningxia Hui Autonomous Region, and the Xinjiang Uygur Autonomous Region. Preoperative endoscopic biopsy confirmed the presence of middle-third or upper third-gastric adenocarcinoma in all study populations treated with surgery. All enrolled patients underwent three-dimensional reconstruction CT scans and other conventional imaging examinations. No patients included in this study had preoperative T4b gastric cancer. Informed consent was obtained from the patients after the study was approved by the ethics committee of the First Affiliated Hospital of Air Force Medical University The distance was also measured in patients who underwent surgery through intraoperative anatomical forceps (fully opened to 2 cm) for comparison with the data measured by three-dimensional imaging. The results were primarily based on the surgical measurements and observations. The patients were divided into concentrated or distributed groups according to the distance. TNM staging was conducted via the eighth version of the AJCC/UICC staging system. In accordance with the Clavien-Dindo classification, an assessment of postoperative complications was conducted. Patients were followed up regularly to compare their survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ① The native place is in Shaanxi Province, Gansu Province, Qinghai Province, Ningxia Hui Autonomous Region, Xinjiang Uygur Autonomous Region;

  * The criteria for patients undergoing laparoscopic radical total gastrectomy include: primary adenocarcinoma of the stomach in the upper third or middle third confirmed by histology; Patients with preoperative diagnosis of clinical T2-T4a (cT2-T4a) gastric cancer were free of tumor invasion of neighboring organs (pancreas, spleen, liver, and transverse colon), paraaortic or splenic hilar lymph node enlargement or fusion, and distant metastases as shown by preoperative abdominal computed tomography (CT), abdominal ultrasound, and endoscopic ultrasound; According to the postoperative pathological diagnosis, total gastrectomy, D2 lymph node resection and radical R0 resection were performed.

Exclusion Criteria:

* ① Patients who did not fully expose the anatomic characteristics of splenic hilar vessels or had evidence of peritoneal spread or distant metastasis during laparoscopic radical gastrectomy;

  * Patients with incomplete clinical data;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient undergoing laparoscopic radical total gastrectomy in the Department of Gastroenterology, Xijing Hospital
Sampling Method: Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 1,3,5 years
  Disease-free survival

SECONDARY OUTCOMES:
The relative position of the splenic artery along the pancreas | Perioperative period
  If the main trunk of the splenic artery runs entirely on the upper surface of the pancreas, it is classified as type I. The type II artery was the middle half of the main splenic artery running inside or behind the pancreas. Similarly, when the distal half of the main splenic artery runs inside or behind the pancreas, it is type III. In addition, if the distal three-quarters or more of the trunk was completely within the pancreas or lay posterior to the pancreas, it was classified as type IV.
Classification of splenic artery branches | Perioperative period
  The splenic artery without branches was categorized as a single-branch type. If two splenic lobe arteries emanate from the terminal, they are defined as two-branch types. Similarly, if the terminal branch has three splenic lobe arteries, it is defined as a 3-branched type; in addition, if there were four or more splenic lobe arteries, it belonged to the multi-branch type.
Overall survival | 1,3,5 years
  Overall survival
The distance between the terminal branch of the splenic artery and the splenic portal | Perioperative period
  If the distance between the bifurcation of the splenic artery and the splenic hilum was less than 2 cm, the patient was assigned to the concentrated group; otherwise, the patient was assigned to the distributed group.
Postoperative complication rate | 30 days
  Postoperative complication rate refers to the frequency or proportion of patients who experience complications following a surgical procedure. This metric is typically calculated over a defined postoperative period, such as within 30 days after surgery. It is an important indicator of surgical safety and the quality of postoperative care. Postoperative complications can vary widely and may include infections, bleeding, organ dysfunction, and other adverse events that affect the patient's recovery and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Li, Study Director — Department of Gastrointestinal Surgery, Xijing Hospital, Fourth Military Medical University
Locations (1):
- The First Affiliated Hospital of PLA Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
After collecting and sorting out the data, share it through the form of article publication or email
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: After collecting and sorting out the data, share it through the form of article publication or email